CLINICAL TRIAL: NCT04031534
Title: Comparative Study of Hypoxia Measured in F-Miso PET/Scan and MRI in Patients With Squamous Cells Carcinoma : Correlation With Immunohistochemistry
Brief Title: Study of Hypoxia Measured in F-Miso PET/Scan and MRI in Patients With Squamous Cells Carcinoma
Acronym: HYPONECK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB16.03
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
Keywords: F-Miso PET scan; Magnetic resonance imaging; immunohistochemistry; Head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measure of hypoxia by F-Miso PET scan and RMI (Experimental): Patient will undergo F-Miso PET scan and MRI to detect hypoxia. Imaging will be correlated with immunohistochemistry on tumour biopsy
  Interventions: Drug: F-Miso PET scan coupled with MRI

INTERVENTIONS:
Drug: F-Miso PET scan coupled with MRI — Patient will undergo F-Miso PET and MRI before surgery for their head and neck cancer. Hypoxia detect with imaging will be correlated with hypoxia detected by immunohistochemistry on tumour biopsy

SUMMARY:
Hypoxia imaging has not been studied extensively by combining PET and MRI data. Few studies performed the double imaging and none associated anatomopathology with it . This study will use a rigorous methodology through the production of PET/MRI images at the same time by transferring the patient directly from PET to MRI. In addition, the population, unlike other studies, will include preoperative patients with 24-hour surgery for hypoxia imaging by obtaining additional data through specific immunohistochemical analysis of hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Patient with squamous cells carcinoma of oropharynx
* Age Superior to 10 years old
* Male or Female
* measurable target according RECIST criteria

Exclusion Criteria:

* -Other histologic cancer than squamous cells carcinoma of oropharynx
* No measurable target
* Presence of metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Comparison of biodistribution of F-Miso PET scan in pre-therapeutic and sequences of MRI in patient with squamous cells carcinoma of oropharynx | 1 year

SECONDARY OUTCOMES:
Correlation of F-Miso PET scan and Magnetic resonance imaging to measure hypoxia | 1 year
Correlation between recurrence free survival at one year and rate of hypoxia determined by the 3 techniques (PET scan, MRI and IHC) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Thureau, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No